CLINICAL TRIAL: NCT06017128
Title: The Effect of Sexual Counseling Based on the PLISSIT Model on Sexual Function, Quality of Life, and Comfort in Patients Undergoing Hip Replacement
Brief Title: Sexual Counseling's Impact on Hip Replacement Patients' Sexual Function and Quality of Life: a PLISSIT Model Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Eda Polat, Research Assisstant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulMU18
Record Dates: First submitted 2023-08-22; First posted 2023-08-30 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hip Arthropathy; Sexual Function Disturbances; Quality of Life
Keywords: Hip Arthropaty; Sexual Function
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Intervention Model Description: This randomized controlled, pre-test-post-test measurement experimental study was designed to determine the impact of sexual counseling based on the PLISSIT model on sexual function, quality of life, and comfort levels in individuals who have undergone total hip replacement surgery.
Masking Description: Individuals will be included in the groups using the randomization method. The randomization of the groups was conducted using the simple-random technique through the use of the website www.random.org.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The experimental group will consist of individuals who will undergo total hip replacement surgery and receive sexual counseling along with an educational booklet.
  Interventions: Other: sexual counseling based on the PLISSIT model
- Control (No Intervention): The control group will be comprised of individuals undergoing total hip replacement surgery without receiving sexual counseling.

INTERVENTIONS:
Other: sexual counseling based on the PLISSIT model — In the initial follow-up, the experimental group will receive information about total hip replacement surgery and its impact on sexual life based on the PLISSIT model. An educational booklet containing information about total hip replacement surgery, the rehabilitation process, and post-operative sexual life will also be prepared and distributed. In the second follow-up (5-7 days after surgery), the experimental group will be provided with information about home care before discharge and returning to sexual life.
  Arms: Intervention

SUMMARY:
This study investigates the influence of sexual counseling using the PLISSIT model on various aspects of patients undergoing hip replacement. The PLISSIT model is employed to guide the counseling process. The research aims to assess how this counseling intervention affects sexual function, quality of life, and overall comfort for these patients. By addressing these factors, the study seeks to shed light on potential improvements in the well-being and experiences of individuals who have undergone hip replacement surgery.

DETAILED DESCRIPTION:
To ensure the proper functioning of the body's systems and the fulfillment of an individual's needs, sufficient movement function is necessary. Decreased movement function, which is crucial for numerous physiological processes, negatively affects overall health status and vital functions. The hip joint is subjected to stress from activities such as walking, running, climbing stairs, lifting weights, and squatting throughout the day. Additionally, conditions like osteoarthritis and rheumatoid arthritis, which emerge with aging, lead to structural and functional abnormalities in the hip joint.

The severe pain and limited movement resulting from issues in the hip joint adversely impact daily life activities, diminishing quality of life. To alleviate pain, improve movement restrictions, and enhance quality of life, Total Hip Arthroplasty (THA) is one of the treatment options. Presently, due to advancements in surgical techniques and materials, THA has become a widely employed method. Literature also indicates increased comfort levels and improved quality of life for individuals after surgery.

One significant component of overall quality of life and general health is a healthy sexual function. Pain and movement limitations in the hip joint also negatively influence individuals' sexual lives. Stiffness, restricted movement, and severe pain in the hip joint lead individuals to be concerned about initiating sexual activity. Studies have shown that after Total Hip Arthroplasty, most patients experience an increase in sexual activity. With the elimination of pain and movement restrictions, individuals engage more comfortably in sexual activities.

However, despite the positive effects of total hip replacement, patients tend to avoid sexual activity due to factors like delayed wound healing, dislocation, joint noises, and uncertainty about resuming sexual relations. Individuals who cannot perform their sexual functions in a healthy manner are negatively affected both physically and psychologically. Moreover, the inability to experience a healthy sexual life, an integral part of marriage and intimate relationships, disrupts the connection between partners. Engaging in sexual activity at the wrong time or in inappropriate positions after surgery can increase the risk of dislocation and reoperation.

Due to all these reasons, the post-operative recovery process and patient comfort are adversely affected. Therefore, in the nursing care provided during the rehabilitation process after total hip replacement, individuals' sexual functions should not be overlooked. Collecting data on patients' sexual functions post-surgery and offering sexual counseling based on their needs are necessary. Detecting and resolving sexual issues are crucial for an effective and expedited post-operative rehabilitation and recovery process. This approach will contribute to the improvement of individuals' physical, social, and psychological health, leading to increased quality of life and comfort levels.

The use of models is highly important in evaluating and resolving individuals' sexual health. The utilization of the PLISSIT model is recommended in providing sexual counseling to healthcare professionals due to its ease of use and systematic approach. The PLISSIT model, developed by Annon in 1976 to guide the resolution of sexual issues, was revised by Taylor and Davis in 2006. The model consists of four stages: P-Permission, LI-Limited Information, SS-Specific Suggestions, and IT-Intensive Therapy.

P (Permission) - Permission: Boundaries for what individuals can and cannot discuss regarding sexuality should be established. In cases where these boundaries are not defined, individuals may not know what they should discuss. In this stage, nurses should allow patients to express their concerns about sexuality and sexual health and encourage them to do so.

LI (Limited Information) - Limited Information: The interventions in this stage aim to inform individuals about sexual matters. This stage involves reviewing the individual's knowledge about sexuality, discussing the effects of the disease and treatments on sexual function, providing information about these effects, and addressing concerns. Providing accurate information helps individuals cope more easily with their concerns about sexuality.

SS (Specific Suggestions) - Specific Suggestions: This stage includes providing individuals/spouses with specific information and recommendations for a more fulfilling sexual life. It is particularly effective for arousal and orgasm disorders and dyspareunia. The recommendations to be made depend on the sexual problem information obtained from the individual. Detailed recommendations such as different positions, interventions, and lubricants can be suggested to individuals with sexual problems.

IT (Intensive Therapy) - Intensive Therapy: This stage is the final stage of the PLISSIT model. If the first three stages of the model are unsuccessful, the intensive therapy stage is employed. The counselor needs to be an expert who has received additional training or should refer the individual to an appropriate unit to provide intensive therapy.

In the literature, it is generally observed that sexual counseling based on the PLISSIT model is provided to women experiencing sexual dysfunction due to reasons such as pregnancy, postpartum, hysterectomy, and mastectomy. Although studies have been conducted worldwide and in our country regarding sexual function after total hip replacement surgery, no study has been found that specifically provides sexual counseling based on the PLISSIT model.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 to 70.
* Willingness to participate in the study.
* Scheduled to undergo hip replacement surgery.
* Being sexually active.
* Ability to engage in verbal communication and being literate.

Exclusion Criteria:

* Having a diagnosed history of a sexual disease in oneself or in one's partner (information about the participant's previous diagnoses will be obtained from the medical team involved in the study).
* Having diagnosed neurological and psychiatric disorders (information about the participant's previous diagnoses will be obtained from the medical team involved in the study).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index | 8 months
  The highest score that can be obtained from the scale is 36 and the lowest score is 2. The cut-off score of the scale is 26.55. Those with a score of 26.55 or less are considered to have female sexual dysfunction. Female Sexual Function Index scores will increase after education according to PLISSIT Model.
International Index of Erectile Function | 8 months
  The severity of erectile function in this area with a maximum score of 30; severe (6-10 points), moderate (11-16 points), mild (17-25 points) and no dysfunction (26 30 points). International Index of Erectile scores will increase after education according to PLISSIT Model.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Tuncer, PhD, Principal Investigator — Istanbul University
Locations (1):
- Prof. Dr. Suleyman Yalcin City Hospital, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researchers will make decisions based on the study outcomes.

REFERENCES:
- [Background] Faghani S, Ghaffari F. Effects of Sexual Rehabilitation Using the PLISSIT Model on Quality of Sexual Life and Sexual Functioning in Post-Mastectomy Breast Cancer Survivors. Asian Pac J Cancer Prev. 2016 Nov 1;17(11):4845-4851. doi: 10.22034/APJCP.2016.17.11.4845. PMID 28030909
- [Background] Issa K, Pierce TP, Brothers A, Festa A, Scillia AJ, Mont MA. Sexual Activity After Total Hip Arthroplasty: A Systematic Review of the Outcomes. J Arthroplasty. 2017 Jan;32(1):336-340. doi: 10.1016/j.arth.2016.07.052. Epub 2016 Aug 11. PMID 27612606
- [Background] Ibrahimoglu O, Gezer N, Ogutlu O, Polat E. The Relationship Between Perioperative Care Quality and Postoperative Comfort Level in Patients With Hip Replacement Surgery. J Perianesth Nurs. 2023 Feb;38(1):69-75. doi: 10.1016/j.jopan.2022.05.068. Epub 2022 Aug 3. PMID 35931599
- [Background] Miettinen HJA, Makirinne-Kallio N, Kroger H, Miettinen SSA. Health-Related Quality of Life after Hip and Knee Arthroplasty Operations. Scand J Surg. 2021 Sep;110(3):427-433. doi: 10.1177/1457496920952232. Epub 2020 Aug 31. PMID 32862793
- [Background] Saray Kilic H, Tastan S. Development of post hip replacement comfort scale. Appl Nurs Res. 2017 Dec;38:169-174. doi: 10.1016/j.apnr.2017.10.004. Epub 2017 Oct 16. PMID 29241512
- [Background] Tuncer M, Oskay UY. Sexual Counseling with the PLISSIT Model: A Systematic Review. J Sex Marital Ther. 2022;48(3):309-318. doi: 10.1080/0092623X.2021.1998270. Epub 2021 Nov 17. PMID 34789082